CLINICAL TRIAL: NCT04584333
Title: Randomised Clinical Trial on the Role of the Dentist in the Control of the Alcoholic Habit, in Elderly Patients with Potentially Malignant Oral Lesions
Brief Title: Role of the Dentist in the Control of the Alcoholic Habit in Patients with Potentially Malignant Oral Lesions
Acronym: ALCODENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PND-2020-ALCODENT
Record Dates: First submitted 2020-09-25; First posted 2020-10-14 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Oral Potentially Malignant Disorders; Alcohol Drinking
Keywords: Alcohol Abuse; Substance Abuse; Monitoring Program; Dentistry; Health Promotion; Clinical trial
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTERVENTION (Experimental): Group 1 (intervention group): depending on the willingness to change evaluated with the RCQ at each visit, the characteristics of the intervention to be performed will be established.
  Interventions: Behavioral: Brief intervention
- NO INTERVENTION (No Intervention): Group 2 (non-intervention group): you will receive the usual information regarding the characteristics of your injuries and the role of tobacco and alcohol in their evolution and the importance of abandoning these habits.

INTERVENTIONS:
Behavioral: Brief intervention — Group 1 (intervention group): depending on the willingness to change evaluated with the RCQ at each visit, the characteristics of the intervention to be performed will be established. Prochaska and DiClemente (1983) proposed a transtheoretical model of change in which different stages of change are identified that have been found to be predictive of adherence to treatment and its efficacy (Prochaska, Norcross and DiClemente, 1994). The RCQ includes three of the stages of change: Precontemplation, Contemplation and Action. In the Precontemplation stage, the person does not consider that he has a problem and has no intention of changing, in the Contemplation stage, he begins to contemplate that he has a problem and the possibility of change is raised and in the action stage, he has already started actively make a change in your behavior.
  Arms: INTERVENTION

SUMMARY:
Introduction: Alcohol is the most consumed psychoactive substance, its consumption is very prevalent and there is a low perception of the risk it poses in our society. Alcohol is a risk factor and a causal factor for multiple pathologies, including cancer and potentially malignant oral lesions (LOPM). The dentist can play a relevant role in the evaluation of consumption, as well as provide brief interventions (BI) to assist them in the cessation of the habit.

Objectives: The main objective is to evaluate the efficacy of the intervention, carried out by dentists, to stop or reduce alcohol consumption in a patient with LOPM.

Material and methods: clinical trial, randomized, with balanced randomization, single-blind (for the evaluator of the results) with 1 experimental arm and a control group, carried out in a single-center manner. Group 1 incident brief intervention and Group 2 no incident intervention (only usual clinical information). 200 patients from the Unit of Oral Medicine, Oral Surgery and Implantology of the University of Santiago de Compostela will participate in this study, they will make an initial visit, one month, three months, six months and one year. In these visits, evaluations related to alcohol consumption, the evolution of injuries, quality of life and satisfaction with the BI were carried out.

Predictable results: If IB contributes to the cessation or reduction of alcohol consumption, and improves the clinical evolution of LOPM, it could be implemented immediately in our Oral Medicine unit and could lay the foundations for its implementation in different public centers and private.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical and histopathological diagnosis of oral lichen planus (OPL) and/or oral leukoplakia (LO) (in all its clinical forms) as chronic LOPMs according to the WHO 2017 classification.
2. Patients over 40 years old
3. Patients in follow-up, with chronic injuries, without medical and/or surgical treatment for at least 1 month
4. Patients with frequent daily alcohol consumption > 1 Standard Beverage Unit (more than two glasses of wine/beer per day or one glass of liquor/distilled drink per day)

Exclusion Criteria:

1. Participants who do not sign the informed consent.
2. Patients with a score above 20 in the AUDIT.
3. Patients undergoing treatment for problems with alcohol and other drugs.
4. Patients with systemic pathology associated with alcohol consumption
5. Pregnant patients.
6. Patients undergoing active pharmacological treatment for OPL.
7. Patients who have undergone surgical resection and/or CO2 laser treatment for LO in the last month.
8. Patients with a history of malignant oral lesions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the intervention | 12 months
  For the main objective, which is to evaluate the efficacy of the intervention, the result will be determined by the percentage of patients who reduce and / or stop the habit in the two arms of the study.

SECONDARY OUTCOMES:
Alcohol consumption | 12 months
  Prevalence and frequency of alcohol consumption in the patients included in the study.The percentages and their distribution will be determined by identifying the number of standard drinking units consumed by the subject on a weekday and weekend.
Alcohol consumption and hazardous alcohol consumption (I) | 12 months
  Prevalence and frequency of alcohol consumption in the patients included in the study It will be determined by means of the AUDIT questionnaire, a self-administered screening test designed by the WHO to assess alcohol consumption. It consists of 10 questions and each question has a series of answers to choose from (score scale from 0 to 4). The eight items of five alternatives score 0 to 4 and the two items (9 and 10) of three alternatives score 0, 2 and 4. The cut-off point of 8 or more indicates the presence of alcohol risk consumption in men, in women 6 and over 20, indicates suspected dependence.
Alcohol consumption and hazardous alcohol consumption (II) | 12 months
  Prevalence and frequency of alcohol consumption in the patients included in the study It will be determined using the CAGE questionnaire originally developed by Ewing and validated in 1974 by Mayfield. It is named after the 4 items it has: C: Cut down; A: Annoyed; G: Guilty; E: Eye opener. It is often used because of its brevity. It is evaluated according to the number of affirmative answers, the greater the dependence. Thus: 0-1: Social drinker; 2: Risk consumption; 3: Harmful consumption; 4: Alcohol dependence
Risky alcohol consumption (GGT) | 12 month
  Quantification of the plasma expression of the GGT markers.GGT (gamma-glutamyl transferase test) which determines the existence of liver damage.It will be analysed in the first visit, after 6 months and a year. Patients will have a sample of peripheral venous blood taken for the study of this marker. To avoid bias in the analysis, all samples will be taken at the Oral Medicine Unit and sent to the same reference laboratory for evaluation and quantification.
Risky alcohol consumption (TDC) | 12 month
  Quantification of the plasma expression of the TDC markers. TDC (tricyclodecane dimethanol, carbohydrate-deficient transferrin) measures a cumulative effect of alcohol consumption, appearing after regular intake of 50-80 g of ethanol per day for at least one week and returning to normal after 15 days of abstinence. It will be analysed in the first visit, after 6 months and a year. Patients will have a sample of peripheral venous blood taken for the study of this marker. To avoid bias in the analysis, all samples will be taken at the Oral Medicine Unit and sent to the same reference laboratory for evaluation and quantification.
Tobacco consumption | 12 month
  The Fagerstrom nicotine dependence test (FTND) will be used (Fagerstrom, 1990). It is one of the most widely used questionnaires for assessing nicotine dependence. It consists of 6 items and has a cut-off point of 6 or more to determine the presence of nicotine dependence.
Evolution of LOPM (I) | 18 months
  Through clinical examination at all visits: stable, worsening or oncological event We will also record the location and size of the lesions.
Evolution of LOPM (II) | 18 months
  We will use the OHIP-14sp (Oral Health Impact Profile - Spanish version), validated by León et al in 2014.A numerical value between 0 and 56 will be obtained, implying that the highest score will represent the greatest effect of oral disorders on the interviewee's quality of life.
Evaluation of the change of stage of readiness to change according to Prochaska and DiClemente. | 18 months
  It will be evaluated by comparing the stages in which the patients are found throughout the follow-up visits.RCQ (Readiness to Change Questionnaire) is an instrument that attempts to measure and operationalize the phase in which patients are in order to modulate the therapeutic intervention by adapting it to the corresponding motivational level. It consists of 12 items and three motivational stages are described (pre-contemplation, contemplation and action). Each stage is represented by 4 items. For each question asked, there are five response options ranging from total disagreement to total agreement. There is a Spanish version validated by Rodriguez-Martos et al that we will use.
Effectiveness of the intrevention | 18 months
  Evaluation of the effectiveness of the brief intervention on alcohol consumption applied by dentists in comparison with the usual advice. The satisfaction questionnaire (CSQ-8) will be used, quantitatively determining the effectiveness.CSQ-8: is a quality evaluation questionnaire for the services provided. Originally published by Atkisson et al., but there is a Spanish version that has been validated. The questionnaire is based on 8 questions to be answered by patients at the end of their stay in the service on a visual analogue scale. Each question is evaluated between 1 and 4 points and satisfaction is directly related to the number of points, so that the sum of these points is a semi-quantitative variable that takes values between 8 and 32 points.This will be done on the last visit to patients in group 1.
Effect of the intervention on the quality of life related to oral health (OHIP) | 18 months
  It will be evaluated by quantitatively comparing the quality of life values at the different stages of monitoring, segmenting the analysis by arm/group and by reduction in consumption.We will use the Oral Health Impact Profile (OHIP) as a measure of people's perception of the social impact of oral disorders on their well-being. To measure oral health-related quality of life, Slade and Spencer in 1994 based themselves on 49 questions known as OHIP-49 , in 1997 Slade developed a short form with 14 questions (OHIP-14) that showed good reliability, validity and accuracy and has been widely used worldwide for various research purposes. This study will use the OHIP-14sp (Oral Health Impact Profile - Spanish version), validated by León et al in 2014.
Effect of the intervention on the quality of life related to oral health (VAS) | 18 months
  It will be evaluated by quantitatively comparing the quality of life values at the different stages of monitoring, segmenting the analysis by arm/group and by reduction in consumption.We will use the VAS ,this is the most widely used scale for measuring pain. It consists of a straight line of 10cm with the words "No Pain" on the left hand side and "The Worst Pain imaginable" on the right hand side and the patient must mark on the line the amount of pain he or she is suffering from. By measuring the distance in centimetres, a figure of 0 to 10 can be deduced. A value of less than 4 in VAS means mild or mild-moderate pain, a value between 4 and 6 implies the presence of moderate-severe pain, and a value of more than 6 implies the presence of very severe pain.
Overall saliva rate (I) | 12 months
  TSG-I (unstimulated). This test is an adaptation of the Schrimer test (a test used to evaluate tear production) and the procedure involves folding the end of the filter paper strip at a right angle before inserting it into the oral cavity under the tongue. When the lips are closed, they come into slight contact with the polyethylene bag. The saliva that collects on the lingual fence during the 5 minutes of the test slowly soaks into the strip. After this time, the strip is removed from the mouth and the result should be read immediately. It will be evaluated on all visits.
Overall saliva rate (II) | 12 months
  TSG-II (stimulated). This test is performed after the TSG-I by applying drops of 4% citric acid solution in the oral cavity.It will be evaluated on all visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Pérez-Sayáns, PhD, Principal Investigator — University of Santiago de Compostela
Locations (1):
- Universidad de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will anonymize and categorize the clinical data of the patients to share the information with the other researchers of the group
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: under request
Access Criteria: under request